CLINICAL TRIAL: NCT01514318
Title: A Long-term Follow Up Study of the Revelation™ Hip Stem
Brief Title: Encore Revelation Hip Stem
Status: Completed | Type: Observational
Sponsor: Encore Medical, L.P. (Industry)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: PS-805
Record Dates: First submitted 2011-12-22; First posted 2012-01-23 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-10

CONDITIONS: Osteoarthritis, Hip; Complications; Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Revelation: Subjects who received the Revelation Hip Stem prior to 2002 and have agreed to come into the office for a single visit.
  Interventions: Device: Revelation Hip Stem (Revelation)

INTERVENTIONS:
Device: Revelation Hip Stem (Revelation) — Subjects who received the Revelation Hip Stem prior to 2002 and still maintain the original device.

SUMMARY:
The purpose of this study is to obtain long-term (10+ yrs) clinical and patient outcomes data on patients who received the Revelation Hip Stem prior to 2002.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have received the Revelation™ Hip Stem as part of a total hip arthroplasty prior to 2002.
* Surgery must have been a primary total hip replacement
* Subject must have received only one primary hip replacement per hospitalization
* Subject must have had a diagnosis of inflammatory tissue disorder, osteoarthritis, post-traumatic arthritis/secondary arthritis or avascular necrosis
* Subject must be willing and able to sign the informed consent document

Exclusion Criteria:

* Subject must not have had any previous hip implants (hemi or total joint)
* Subject has a mental condition that may interfere with the ability to give an informed consent (i.e., severe mental retardation such that the subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Subject is a prisoner
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include only subjects who received the Revelation Hip Stem prior to 2002 and who voluntarily consent to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frosty Moore, M.D., Principal Investigator — Westlake Orthopaedics Spine & Sports
Locations (1):
- Westlake Orthopaedics Spine & Sports, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The site had a list of patients to call based on previous enrollment into an IDE study from back in 1998. There was not additional recruitment required.
Pre-assignment Details: Assignment was based on subjects signing the consent form. They were either in the study or not.
Period: Overall Study
Arm/Group | Revelation
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Revelation
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 61.6 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Survivorship of the Device
Description: The subject meets the inclusion/exclusion criteria of the study and received a Revelation Hip Stem prior to 2002 that has survived intact without any type of surgery to revise or remove parts or the whole prosthesis.
Time Frame: 10 year
Population: Subjects who signed the consent form and completed the study paperwork.
Measure: Number; unit: participants
Arm/Group | Revelation
Number analyzed (Participants) | 8
participants | 8

2. Secondary Outcome: Western Ontario McMaster Arthritis Index (WOMAC)
Description: Standardized questionnaire used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip. It assesses the pain, joint stiffness, physical, social & emotional function of a person with osteoarthritis in determining the overall level of disability. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). For each item, the possible range of scores is therefore 0-100. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in and out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties.
Time Frame: 10 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Revelation
Number analyzed (Participants) | 8
units on a scale | 17.4 (4.6)

3. Secondary Outcome: Harris Hip Score
Description: A tool for the evaluation of how a patient is doing after their hip is replaced. Based on a total of 100 points possible, each question is awarded a certain number of points based on how it is answered. Questions are further grouped into four categories. The first category is pain, the second category is function, third is functional activities and finally the physical exam results are tabulated, and based on your range of motion. The score is reported as 90-100 for excellent results, 80-90 being good, 70-79 fair, 60-69 poor, and below 60 a failed result.
Time Frame: 10 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Revelation
Number analyzed (Participants) | 8
units on a scale | 82.4 (15.4)

ADVERSE EVENTS:
Arm/Group | Revelation
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Small patient population to choose from and difficulty in locating people who have not been seen by the doctor in almost 10 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less